CLINICAL TRIAL: NCT03951155
Title: Effectiveness of Relaxation Technique (Muscle Relaxation) for Behavioral Management of ADHD Children During Dental Treatment. (Randomized Clinical Trial)
Brief Title: Effectiveness of Relaxation Technique for Behavioral Management of ADHD Children During Dental Treatment.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nouran Khalifa Hamed, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14422016457337
Record Dates: First submitted 2019-05-11; First posted 2019-05-15 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; behavioral management; dental management
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Muscle Relaxation; Relaxation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor responsible for evaluating child behavior & cooperation will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADHD Group (Experimental): Muscle Relaxation technique for behavioral management
  Interventions: Behavioral: Muscle Relaxation
- Tell Show Do Group (No Intervention): Tell Show Do Technique for behavioral management

INTERVENTIONS:
Behavioral: Muscle Relaxation — * Ask the child to lie down in a comfortable position. Ask him/her to notice how their muscles feel in each part of the body. Taking one area of the body at a time (face, shoulders, arms, hands, fingers, abdomen, legs, feet, and toes).
  * Instruct the child to contract the muscles for 5 seconds, take a deep breath, and release.
  * Next, instruct the child to contract all muscles simultaneously, hold for 5 seconds, then release.
  * Finally, ask him/her to notice how his/her muscles feel after the exercise.
  Other Names: Relaxation technique
  Arms: ADHD Group

SUMMARY:
Evaluation of effect of relaxation technique (Muscle Relaxation) on behavioral management and anxiety control of ADHD children during dental treatment.

DETAILED DESCRIPTION:
Evaluation of effect of relaxation technique (Muscle Relaxation) on behavioral management and anxiety control of ADHD children during dental treatment compared to Tell Show Do technique (control group) using modified Frankl scale.

ELIGIBILITY:
Inclusion Criteria:

* Children: 6 to 9 years old ADHD children
* Teeth: Teeth requiring dental treatment or preventive measure.

Exclusion Criteria:

* Non ADHD children.
* ADHD children having allergy to local anaesthesia or systemic problem that contraindicate dental treatment.
* Refusal of participation

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Modified Frankl Scale for child cooperation | one day
  Rating 1: DEFINITLY NEGATIVE (--): Refusal of treatment, crying forcefully, fearful, or any other overt evidence of extreme negativism.
  * Rating 2: NEGATIVE (-): Reluctant to accept treatment, uncooperative, some evidence of negative attitude but not pronounced, i.e. sullen, withdrawn.
  * Rating 3: NEGATIVE POSITIVE (-+): Fluctuation between uncooperativeness and some evidence of unpronounced negative attitude, and cautious acceptance to treatment with reservation shifting throughout the visit.
  * Rating 4: POSITIVE (+): Acceptance of treatment; at times cautious, willingness to comply with the dentist, at times with reservation but patient follows the dentist's directions cooperatively.
  * Rating 5: DEFINITLY POSITIVE (++): Good rapport with the dentist, interested in the dental procedures, laughing and enjoying the situation.

SECONDARY OUTCOMES:
Completion of treatment | one day
  weather the dental treatment completed or not

IPD SHARING:
Plan to Share IPD: No
All data, information, participant's personal information, family history, social and medical history will be stored in the files assigned to each patient with limited access to minimum number of individuals necessary for quality control, audit, and analysis.